CLINICAL TRIAL: NCT03917277
Title: Musculoskeletal Ultrasound of the Ankles in Erysipelas-like Erythema of Familial Mediterranean Fever
Acronym: ECHOPERY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190233
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Erysipelas
Keywords: Erysipelas-like erythema; Familial Mediterranean Fever; Musculoskeletal ultrasound
MeSH Terms: conditions — Erysipelas; Familial Mediterranean Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musculoskeletal ultrasound of the ankle (Experimental): see "Intervention description"
  Interventions: Device: Musculoskeletal ultrasound

INTERVENTIONS:
Device: Musculoskeletal ultrasound — Ankle sonographic examination will be performed using Samsung UGEO H60 ultrasound machine in use since 2016. In order to optimize reproducibility, all examinations will be performed by a single examiner. Multiplanar (longitudinal/transverse) scanning will be done in B- and PD-mode to identify pathologies defined by the OMERACT network in the following structures:
  1. Talocrural joint:synovial fluid (scored 0-3);synovitis with synovial hypertrophy and PD signal (each scored 0-3); bone erosion with distance between cortices and presence/absence of DP signal
  2. Tibialis anterior,tibialis posterior, extensor digitorum longus, fibularis brevis,fibularis tertius,and calcaneal tendons: presence/absence of tenosynovitis, thickening, hypoechogenicity, nodularity, fusiform aspect, and DP signal
  3. Calcaneal enthesis: presence/absence of thickening,hypoechogenicity,calcification, cortical irregularity,and DP signal
  4. Retrocalcaneal and calcaneal bursa: presence/absence of bursitis and DP signal

SUMMARY:
Erysipelas-like erythema (ELE) and arthritis are common manifestations affecting the ankle in Familial Mediterranean Fever. Musculoskeletal ultrasound examination of the ankle has never been performed during an episode of ELE. We hypothesize that ELE is associated with underlying musculoskeletal pathology. In order to support this hypothesis, ankle musculoskeletal ultrasound will be performed within 24 hours of onset of ELE in 15 patients diagnosed with FMF. Results will be correlated with clinical parameters, serum inflammatory markers, and ankle radiography.

DETAILED DESCRIPTION:
Erysipelas-like erythema (ELE) is the pathognomonic cutaneous manifestation of familial Mediterranean fever (FMF). It typically presents with painful, well-demarcated, and unilateral erythema overlying the ankle, and resolves spontaneously within 24 to 72 hours. Its incidence varies from 1% to 48% in the literature, depending on gender and ethnicity. Joint involvement during FMF is more common than ELE, affecting between 17% and 77% of patients. It is most often monoarticular and involves the ankles in almost half of cases. Concomitant ELE is described in up to 43% of patients. However, the overlap between the clinical presentation of ELE and ankle arthritis in FMF poses a diagnostic challenge.

Musculoskeletal ultrasound is a simple and sensitive technique for the evaluation of articular and peri-articular structures. Only one study described sonographic articular involvement in FMF. In 29 asymptomatic patients, an increased prevalence of knee effusion, retrocalcaneal bursitis and medial tenosynovitis of the ankle was noted compared with the control group. Irrespective of joint involvement, an increased prevalence of enthesopathy has also been documented by ultrasound in patients with FMF, thus strengthening its association with spondyloarthropathy. However, no study has evaluated by ultrasound the articular and peri-articular involvement of the ankle during an episode of ELE. To date, the treatment of ELE involves ankle offloading and administration of analgesics. By allowing a better understanding of its pathogenesis, sonographic confirmation of articular and peri-articular involvement of the ankle during an episode of ELE will potentially allow to optimize its therapeutic management.

The study population involves over 600 patients with FMF followed at Tenon Hospital, which is part of the French Reference center for rare auto-inflammatory diseases and amyloidosis (CEREMAIA). Eligible patients will be contacted by mail or email to inform them of the study. Those interested in participating will be advised to contact the investigators by email or phone at the onset of ELE. Patients presenting with ELE during their visit in the internal medicine department of Tenon Hospital will also be screened for eligibility.

A visit between the participant and attending physician will be scheduled within 24 hours of the onset of ELE. The usual management of ELE will not be altered. The visit will include a questionnaire and physical examination to assess the presence of typical manifestations of FMF attacks, such as chest and/or abdominal pain, as well as to exclude systemic toxicity in favor of an alternative infectious diagnosis. It will involve a blood test for complete blood count and C-reactive protein measurement to confirm the inflammatory syndrome, as well as an x-ray of the ankles to exclude an underlying structural pathology. Analgesics will be prescribed for symptomatic relief. The patient will be advised to go the emergency room if ELE and/or fever persist beyond 72 hours, or if symptoms suggestive of an infectious process develop (significant worsening of general state, cardiorespiratory symptoms, pre-syncope or syncope, etc).

The inclusion visit for the study will be integrated to this medical consultation. Once free and informed consent is obtained, the following clinical data will be collected: age, sex, weight, height, body mass index, ethnicity, age at onset of FMF symptoms, age at diagnosis of FMF, genotype, frequency of attacks, diagnosis of amyloidosis, spondyloarthropathy, inflammatory bowel disease and/or vasculitis, previous episodes of ankle arthritis, duration and location of ELE at inclusion, total duration of ELE, presence of fever, serositis and/or myalgia, and current treatment for FMF. In search of potential confounding factors for sonographic musculoskeletal abnormalities, the following data will also be collected: professional occupation, physical activity (type and frequency), presence of pes planus or cavus, pre-existing ankle pain, and chronic ankle edema. Sonographic evaluation of the articular and periarticular structures of the two ankles will be performed using the Samsung UGEO H60 echograph, in operation since 2016. In order to ensure reproducibility, the evaluation will be completed by a single examiner throughout the study.

Following the inclusion visit, a follow-up by email or phone will be done within one week of inclusion in order to confirm the exact duration of ELE. This information will allow us to confirm the diagnosis of ELE, which normally resolves spontaneously within 72 hours, in contrast to its main differential diagnosis, namely erysipelas. Thereafter, there will be no additional follow-up as part of this study.

The patient inclusion phase will last 8 months, followed by 3 months of data analysis. We estimate that 8 months will be sufficient to recruit 15 patients among our study population. The number 15 was arbitrarily chosen because FMF is a rare disease, and the incidence of ELE in this population is highly variable and therefore poorly defined in the literature.

Regarding data analysis, clinical, biological, radiographic and sonographic data will be presented as medians (± interquartile interval) when these are continuous variables, and as absolute numbers with proportion when these are categorical variables. Sonographic and radiographic findings will be compared between the ankles ipsilateral and contralateral to ELE. Continuous variables will be compared with the Mann-Whitney test. Categorical variables will be compared with the Fisher test. In order to determine whether clinical and paraclinical parameters are correlated with the presence of sonographic musculoskeletal pathologies, univariate and multivariate analyses will be performed using a logistic regression model. A p value ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient followed by the National reference center for autoinflammatory diseases and inflammatory amyloidosis (CeRéMAIA) at Tenon Hospital in Paris
* Patient with a diagnosis of FMF based on Livneh criteria and supported by 2 pathogenic MEFV mutations
* Patient with unilateral ankle ELE for less than 24 hours and whose diagnosis is confirmed a posteriori by its spontaneous resolution in 72 hours
* Patient affiliated or entitled to an affiliation to a social security system
* Provision of informed consent

Exclusion Criteria:

* Incapacity to answer questions, express him(her)self clearly, or collaborate with the performance of the musculoskeletal ultrasound
* Previous surgery, significant trauma, destructive arthropathy, and any other pathology affecting the musculoskeletal structures of the ankle and thus influencing its sonographic examination
* Previous diagnosis of gout
* Current pregnancy
* Patient deprived of liberty or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal ultrasound evaluation of the ankle | Within 24 hours of the onset of ELE
  Presence of one or more of the following musculoskeletal pathologies identified by sonographic examination of the ankle: synovial fluid, synovitis, and/or bone erosions in the talocrural joint; tendinous anomalies in the tibialis anterior, tibialis posterior, extensor digitorum longus, fibularis brevis, fibularis tertius, and calcaneal tendons; calcaneal enthesopathy, and retrocalcaneal and calcaneal bursitis.

SECONDARY OUTCOMES:
Comparison of sonographic and radiographic findings between both ankles | Within 24 hours of the onset of ELE
  Compare findings on musculoskeletal ultrasound and radiography between the ankle ipsilateral and contralateral to ELE.
Sonographic evaluation of soft tissue thickness of the ankle | Within 24 hours of the onset of ELE
  Measure and compare soft tissue thickness between the ankle ipsilateral and contralateral to ELE
Correlation of sonographic findings with patients' characteristics | Within 24 hours of the onset of ELE
  Correlate presence of musculoskeletal ultrasound pathologies of the ankle ipsilateral to ELE with clinical and paraclinical parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie GEORGIN-LAVIALLE, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Karine LOUATI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Interne, Paris, France